CLINICAL TRIAL: NCT06971679
Title: INVESTIGATING THE EFFECT OF FLIPPED CLASSROOM METHODS COMBINED WITH PROBLEM-BASED LEARNING ON NURSING STUDENTS' KNOWLEDGE AND ATTITUDES REGARDING PATIENT SAFETY
Brief Title: FLIPPED CLASSROOM METHODS COMBINED WITH PROBLEM-BASED LEARNING ON NURSING STUDENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gülcan Karabulut (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor-Investigator, Gülcan Karabulut, Research Assistant, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TBAEK-701
Record Dates: First submitted 2025-04-20; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: PROBLEM-BASED LEARNING; NURSING STUDENTS; FLIPPED CLASSROOM METHODS; PATIENT SAFETY
Keywords: Problem-based learning; Nursing students; Flipped Classroom Methods; Patient Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Didactic Group (No Intervention): In the first week of the clinical practice, the control group students were given patient safety training by the researcher using the classical didactic method on the same day and time as the intervention group students. After the training, a case test was applied to the students.
- Flipped Group (Experimental): In the first week of the clinical practice, the E-learning module prepared by the researchers within the scope of the flipped education method was shared with the intervention group students and all students were shown in a conference room. After the training, PBL modules (different cases related to patient safety for each group) were shared with the students divided into groups of 3-5 students within the scope of PBL and they were given one week to prepare. In the other weeks of the clinical practice, face-to-face case discussions were held with the groups. These case discussions lasted an average of 40 minutes.
  Interventions: Behavioral: Flipped Method

INTERVENTIONS:
Behavioral: Flipped Method — In the first week of the clinical practice, the E-learning module prepared by the researchers within the scope of the flipped education method was shared with the intervention group students and all students were shown in a conference room. After the training, PBL modules (different cases related to patient safety for each group) were shared with the students divided into groups of 3-5 students within the scope of PBL and they were given one week to prepare. In the other weeks of the clinical practice, face-to-face case discussions were held with the groups. These case discussions lasted an average of 40 minutes.
  Arms: Flipped Group

SUMMARY:
Nurses need to develop critical thinking skills to be competent in flexible, personalized, and situation-specific problem solving in today's healthcare environment of rapid change and increasing information. This means that nursing education should prepare nursing students to meet the needs of patients, serve as leaders, develop scientific rigor for the benefit of patients, and make decisions based on critical thinking. In addition to transferring theoretical knowledge, nursing education is also very important in terms of putting students' knowledge into practice and improving students' comprehensive qualifications.

DETAILED DESCRIPTION:
One of these qualities is the fundamental responsibility of nurses to ensure patient safety. It is estimated that 421 million hospitalizations occur every year in the world. Approximately 7.42 million adverse events occur during these hospitalizations, and patient harm is the 14th leading cause of global mortality. Many universities are looking for teaching methods that can improve students' clinical decision-making abilities and self-directed learning in order to provide safe and quality nursing care. Lack of patient safety knowledge is one of the educational problems of nursing students leading to unsafe practices.Early education on patient safety is crucial in preparing nurses to be competent in patient care. Therefore, offering patient safety education courses at the undergraduate level using an innovative approach is important to improve patient safety and quality in nursing care.

Various innovative approaches are used in nursing education to improve students' critical thinking and problem-solving skills. These include team-based learning, concept mapping, case studies and problem-based learning (PBL) and flipped classroom model. In the flipped classroom model, students are presented with course materials prior to class and then class time is spent gaining in-depth understanding through interactive activities. Studies have shown that the flipped classroom model improves students' academic performance and satisfaction. However, compared to traditional lecture-based classes, reverse classes have been reported to be more effective in improving academic performance and course evaluation as well as developing engagement and higher-order thinking skills in nursing students. Problem-based learning (PBL), one of the important teaching methods that improve nursing students' clinical performance and critical thinking skills, can be used as an in-class activity in flipped classrooms. However, some studies indicate that the simple implementation of PBL instruction can challenge students' systematic understanding of the required knowledge and that this model is more difficult for students with low learning ability and performance, resulting in learning fatigue and worse learning outcomes than expected. Several studies have explored the combined use of reverse classrooms and PBL in nursing education. However, it is important to investigate how to maximize the impact of pre-course self-study to promote the development of students' abilities. Therefore, this study aims to determine the effect of patient safety education provided by combining the flipped classroom model with problem-based learning within the scope of nursing management course on nursing students' patient safety knowledge, attitudes and perceptions.

ELIGIBILITY:
Inclusion Criteria:

* 2024-2025 Academic Year Fall Semester enrolled in the Nursing Management Lesson,
* agreed to participate in the study
* completed the data collection forms completely

Exclusion Criteria:

* want to leave the research at any time of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Socio-demographic Characteristics Form | Baseline
  The socio-demographic characteristics form prepared by the researchers consisted of four questions: age, gender, the status of receiving training on medical errors and patient safety outside the curriculum, and the source of the training.
H-PEPSS TR | Baseline and 4 weeks after the intervention
  The H-PEPSS TR is a 23-item, two-level measurement tool. It consists of two main dimensions: "Classroom" and "Clinical environment". The scale consists of six sub-dimensions. Item total score averages are used in the whole scale and sub-dimensions. Each item of the scale is evaluated as "Strongly disagree-1 point" and "Strongly agree-5 points" on a five-point. The higher the score obtained from the "classroom" dimension and sub-dimensions of the scale, the higher the participants' perceptions of patient safety knowledge developed in the classroom environment.The higher the score obtained from the "clinical environment" dimension and sub-dimensions of the scale, the higher the participants' perceptions of patient safety competence developed in the clinical environment.
Patient Safety Competency Self-Assessment Tool | Baseline and 4 weeks after the intervention
  Item total score averages are used in the total scale and sub-dimensions. The minimum score that can be obtained from the scale and sub-dimensions is 1 and the maximum score is 5. Higher mean scores indicate that students have better knowledge, skills and attitudinal competencies in patient safety. Since the instrument is a multidimensional scale, the mean scores of the total scale, 3 dimensions and 12 factors are evaluated separately. Each item of the scale is evaluated in a five-point Likert scale with different expressions in each dimension; The knowledge dimension consists of 2 factors and 6 items in total. Its evaluation is as "1=I have no knowledge at all, 5=I know very well". The skills dimension consists of a total of 6 factors and 21 items. Its evaluation is as "1=I cannot do it at all, 5=I can do it very easily". Attitude dimension consists of 4 factors and 14 items. The evaluation is "1=Strongly disagree, 5=Strongly agree".
Case Test and Open-Ended Question | 4 weeks after the intervention
  A 20-question patient safety events test and two open-ended case questions (cause of error, risks, influencing factors, developing strategies for prevention, incident reporting and root causes) were created by the researchers and administered as a test. The test was evaluated out of 100 points.
  This is an evalution test exam, the minimum point is 65 for success.
PBL Modules | 4 weeks after the intervention
  Modules were prepared by the researchers. The cases and questions in the case test were structured as PBL cases to compare the module content assessments. In PBL modules, students were asked to conduct root cause analysis on reported medical error scenarios. In this analysis, module work including the cause of the error, risks, influencing factors, suggestions for prevention, extraction of the root causes of the event, etc. was carried out. In the evaluation of each group, points were given according to the 100-point system. Case test results were evaluated as correct answers. PBL cases were scored on the realization of the implementation steps.
  This is an evaluation exam and 65 point for be success.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Kumluca Faculty of Health Science, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided